CLINICAL TRIAL: NCT06398327
Title: Efficacy Of Proinflammatory Cytokines in the Clinical And Radiographic Outcomes of Different Primary Molar Pulpotomy Agents: A Comparative Study Featuring A Novel Biomarker For Pulpal Diagnosis
Brief Title: Efficacy Of Proinflammatory Cytokines in The Primary Molar Pulpotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, AYBİKE BAŞ, assisstant proffessor- pediatric dentistry, Ataturk University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: B.30.2.ATA.0.01.00/345
Record Dates: First submitted 2024-04-07; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Pulp Disease, Dental
Keywords: Presepsin; MTA; Neo MTA; Biodentine; zinc oxide eugenol; ıl-6; IL-8; Pulpal inflammation; Pulpotomy treatment; Primary molar teeth
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Zinc oxide eugenol cement (Active Comparator): During pulpotomy treatment, a blood sample was taken from the coronal pulp and stored. The remaining pulp tissue was covered with ZOE, randomly selected from among four material groups. The teeth treated with ZOE were monitored for 12 months. Subsequently, the levels of IL-6, IL-8, and Presepsin in the blood were measured using the ELISA method and noted in ng/ml. Thus, the effect of the material used on the success of the treatment was determined based on the level of pulpal inflammation before treatment.
  Interventions: Procedure: PULPOTOMY TREATMENT
- Mineral Trioxide Aggregate (MTA) (Active Comparator): During pulpotomy treatment, a blood sample was taken from the coronal pulp and stored. The remaining pulp tissue was covered with MTA, randomly selected from among four material groups. The teeth treated with MTA were monitored for 12 months. Subsequently, the levels of IL-6, IL-8, and Presepsin in the blood were measured using the ELISA method and noted in ng/ml. Thus, the effect of the material used on the success of the treatment was determined based on the level of pulpal inflammation before treatment.
  Interventions: Procedure: PULPOTOMY TREATMENT
- NeoMTA (newly developed mta) (Active Comparator): During pulpotomy treatment, a blood sample was taken from the coronal pulp and stored. The remaining pulp tissue was covered with NeoMTA, randomly selected from among four material groups. The teeth treated with NeoMTA were monitored for 12 months. Subsequently, the levels of IL-6, IL-8, and Presepsin in the blood were measured using the ELISA method and noted in ng/ml. Thus, the effect of the material used on the success of the treatment was determined based on the level of pulpal inflammation before treatment.
  Interventions: Procedure: PULPOTOMY TREATMENT
- Biodentine (biomaterial) (Active Comparator): During pulpotomy treatment, a blood sample was taken from the coronal pulp and stored. The remaining pulp tissue was covered with Biodentine, randomly selected from among four material groups. The teeth treated with Biodentine were monitored for 12 months. Subsequently, the levels of IL-6, IL-8, and Presepsin in the blood were measured using the ELISA method and noted in ng/ml. Thus, the effect of the material used on the success of the treatment was determined based on the level of pulpal inflammation before treatment.
  Interventions: Procedure: PULPOTOMY TREATMENT

INTERVENTIONS:
Procedure: PULPOTOMY TREATMENT — During pulpotomy treatment, a bleeding sample was taken from the pulp and levels of presepsin, IL-6 and IL-8, which are important inflammation markers, were determined. During the treatment, MTA, Neo MTA, Biodentine and ZOE groups were randomly selected and the remaining pulp tissue was covered. After pulpotomy treatment, the teeth were followed for one year. Treatment success was evaluated according to the material used in teeth with high levels of inflammation at the beginning.

SUMMARY:
One of the main goals of pediatric dentistry is to preserve the functions and structures of primary teeth until the time of exfoliation. Especially carious lesions are the main factor in the early loss of primary teeth. Today, primary teeth can be kept in the mouth by applying different treatments depending on the degree of inflammation caused by carious lesions in the pulp tissue.Coronal pulpotomy application in asymptomatic primary teeth with deep carious lesions near the pulp is one of the most common methods to achieve the goal of retaining the tooth in place. The purpose of the pulpotomy technique is to remove the affected pulp tissue and maintain the normal function of the unaffected root pulp tissue until the tooth is naturally ready to exfoliate.

Studies have shown that the degree of pulp inflammation and the materials used are effective in the success of this treatment. In studies evaluating pulpal inflammation, many biomarkers have been shown to play significant roles at different levels of inflammation. Recently, Presepsin has been studied as a biomarker for detecting bacterial infections. However, there is no study in the literature on the use of Presepsin as a biomarker in endodontic treatments. In our study, it is thought that Presepsin biomarker could be detected in cases of acute or chronic infection in pulp tissue and could be considered as one of the mediators of pulpal inflammation.

Based on this, the aim of our study is to investigate whether the materials used in covering the pulp or the level of inflammation in the remaining pulp tissue is more important for the success of pulpotomy treatment. The inflammation level in the remaining pulp tissue will be measured using IL-6, IL-8, and Presepsin. Then, the one-year success of treatment in different groups where pulp tissue is randomly covered with MTA, NeoMTA, Biodentine, and Zinc oxide eugenol will be demonstrated. Thus, it will be evaluated whether materials previously found to be quite successful in other studies achieve success in pulps with high inflammation levels.

DETAILED DESCRIPTION:
Tooth decay is a commonly encountered chronic infectious disease in children. Coronary pulpotomy treatment is generally preferred for teeth with deep decay lesions that are clinically and radiographically asymptomatic. The success of this treatment method is highly dependent on the inflammatory status of the pulp and the materials used. In predicting the clinical success of pulpotomy treatment, the severity of pulp inflammation must also be evaluated. A molecular approach that aids in the clinical distinction between reversible and irreversible pulpitis can increase the success rate of vital pulp therapy by accurately assessing the inflammation status of the pulp. Although various mediators' increases in advanced pulpal inflammation have been examined in many previous studies, the role of many biomolecules involved in pulpal inflammation has not yet been determined. Due to the complex nature of inflammatory pulp disease, it is unlikely that a small number of mediators would provide sufficient information to diagnose advanced inflammatory disease. Therefore, studies aimed at identifying new mediators remain relevant in dentistry. Presepsin, discovered in 2004, is a biomarker with high sensitivity and specificity that is highly important in the early diagnosis of bacterial diseases in medicine. When dental literature is reviewed, it is observed that presepsin has not been evaluated for the detection of bacterial inflammation in the pulp, and it is believed that this biomarker could be used for the early detection of pulpal inflammation. Thus, with the ability to measure presepsin levels using patient kits, pulpal inflammation can be quantitatively evaluated, aiding in the provision of accurate pulp treatments.The aim of our research is to investigate whether presepsin, a new biomarker that can be rapidly detected in bacterial infections, can also be used as a mediator in the detection of pulpal infections, and to evaluate the levels of the reliable markers of pulpal inflammation, IL-8 and IL-6, comparing the effect of these mediators on the success of treatment with the most successful materials used in pulpotomy treatment, MTA, Neo MTA, Biodentine and Zinc oxide eugenol.

This study was conducted in accordance with the Ataturk University Faculty of Medicine Ethics Committee approval (Date: 05.2021/ Session no:04/ Decision no:66) and guidelines of the Helsinki Declaration. Also the parents of child patients were comprehensively briefed about the procedures before the treatment and their written consents were obtained. Initially, a total of 75 children aged 4-9 years old (36 girls and 39 boys) with no systemic disease and presenting at least one primary second molar indicated for pulpotomy were included in the study and 4 pulpotomy agents (MTA, Biodentine™, NeoMTA™ and ZOE) were randomly divided into four study groups of 30 teeth and pulpotomy was applied to a total of 120 teeth.

In order to randomly distribute the study groups, Research Randomizer (Version 4.0) computer software from http://www.randomizer.org/ was used to generate a list before starting pulpotomy and pulpotomy agents were used accordingly.

Protocols for Treatment and Sample Storage:

For a better visibility a rubber-dam is placed over the tooth requiring pulpotomy following local anesthesia. Endodontic cavity was accessed by first removing the carious tissue, unroofing the pulp chamber with diamond round bur (no:18), removing the coronal tissue using a sterile tungsten carbide round bur (no:14) mounted low-speed contra-angled handpiece and clearing the remaining pulpal tissue with an excavator.

Before managing the pulpal hemorrhage, a sterile cotton pellet was placed over the pulp tissue for 30-45 sec. in order to obtain pulpal blood samples and specimens were collected into heparin coated tubes (Vacutainer, BD,USA) with 1mg saline solution and they were stored at -20 oC (-4.0°F) for 6 months until the day of testing.

Then pulpal hemostasis was achieved by placing 0.5 % NaOCl over the canal orifices for 30 sec. Primary molars, in which pulpal hemorrhage was controlled were randomly assigned to 4 different study groups (ProRoot MTA, Biodentine™, NeoMTA™, and ZOE respectively) and they were treated with pulpotomy. Glass ionomer cement was applied over all pulpotomy medications used in the study and pulpotomized teeth were restored with stainless steel crowns (SSCs).

Thawing Process and Assessment:

Samples were thawed at room temperature and centrifuged at 4000 rpm for 15 min. Then cotton pellets were removed from the test tubes and levels of presepsin, IL-6 and IL-8 were measured using enzyme-linked immunoassay (ELISA) [Human presepsin ELISA kit (Cat.No:E3754Hu, BT LAB,China),Human IL-6 ELISA Kit (Cat.No:E0090Hu,BT LAB,China), Human IL-8 ELISA Kit (Cat.No:E0089Hu, BT LAB,China)] test in accordance with the manufacturer's instructions. Kit measurement ranges for presepsin, IL-6 and IL-8 were 5-1000ng/L, 2-600ng/L and 5-1000ng/L respectively. The inter- assay CV were <10% for all biomarkers.

Clinical & Radiographic Assessment Method:

Primary second molars were assessed clinically and radiographically at the post- treatment 6th and 12th months.

Spontaneous or stimulated pain, swellings in vestibular sulcus, fistula, pathological mobility, sensitivity to percussion and palpation, regional lymphadenopathy adjacent to the pulpotomized teeth were clinically assessed and presence of any of these symptoms were regarded as failed pulpotomy.

Radiolucency in the periapical or furcation areas, internal and external root resorptions, calcified root canals, widened periodontal ligament were radiographically evaluated and presence of any of these symptoms were also regarded as failure.

Additionally, presence of lesions in periapical or furcation areas in radiographs were also accepted as failure and these teeth underwent root canal treatment or extraction. Furthermore, teeth with internal root resorption were regarded as radiographically failed and they were just followed-up until any symptom occurred.

Statistical Analysis Descriptive statistics (count, ratio, mean, standard deviation, minimum and maximum variables) were used to summarize the set of data in the present study. Fisher's exact test was employed to analyze the relationship between pre-treatment clinical findings and dental pathologies developed at the post-treatment 12th month when pathologies became more apparent. Relationship between the mean levels of pulpal inflammatory biomarkers and dental pathologies occurred at the post-treatment 12th month was analyzed using Mann-Whitney U test. Mann-Whitney U test was also used to compare the mean levels of inflammatory biomarkers and clinical findings. Kruskal Wallis test was used to compare the differences between the mean scores of inflammatory biomarkers by the pulpotomy agents used.

Threshold values were calculated with Receiver Operating Characteristics (ROC) analysis and then these obtained values were used to determine the highest biomarker scores in the pulpotomy material groups. All study analysis were performed with IBM® SPSS® Statistics 25 at a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children between the ages of 6-9
2. Children who do not have any systemic disease
3. Primary second premolars in which physiological root resorption has not started.
4. Cases where tooth decay at the interfaces exceeds ½ of the dentin thickness.
5. Primary second premolars with provoked pain

4. Lack of percussion sensitivity 5. Absence of radiolucent image in the periapical and furcal areas on x-ray 6. Clinical absence of abscess and fistula

Exclusion Criteria:

1. Children with systemic diseases
2. Having percussion sensitivity
3. Radiolucent appearance in the periapical and furcal areas on x-ray
4. Clinical presence of fistula
5. Having night pain

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Clinical Success After Pulpotomy Treatment | 6 Month - 1 Year
  No signs of abscess or any swelling related to the tooth, no signs of fistula or other pathology, no signs of pathologic mobility, no post-operative pain, no pain on palpation or percussion of the tooth.
Radiographic Success After Pulpotomy Treatment | 6 Month - 1 Year
  No signs of root resorption (internal or external), no signs of furcation involvement or periapical radiolucency, no signs of loss of lamina dura, presence of normal appearance of periodontal ligament space.
IL-6 amount measurement using ELISA kit | 6 Month - 1 Year
  IL-6 levels were measured in ng/ml using the ELISA method. The measurement procedure was followed according to the manufacturer's instructions. The anti-IL-6 polyclonal antibody was pre-coated on 96-well plates. Blood samples and a biotin-conjugated antibody were added to the wells supplemented with Avidin-Biotin-Peroxidase Complex and 3,3',5,5'-tetramethylbenzidine in a mildly acidic buffer. A blue-colored product was produced and turned to yellow after an acidic stop solution was added. The intensity of the color yellow was proportional to the IL-6 amount bound on the plate. The optical density absorbance was measured spectrophotometrically at 450nm in a microplate reader and the concentration of IL-6 was calculated. For the expression of IL-6 concentrations in the samples, a standard curve was used.Optimal threshold values (cut-offs) for biomarkers were determined based on sensitivity and specificity, which were calculated from a ROC curve.
IL-8 amount measurement using ELISA kit | 6 Month - 1 Year
  IL-8 levels were measured in ng/ml using the ELISA method. The measurement procedure was followed according to the manufacturer's instructions. The anti-IL-8 polyclonal antibody was pre-coated on 96-well plates. Blood samples and a biotin-conjugated antibody were added to the wells supplemented with Avidin-Biotin-Peroxidase Complex and 3,3',5,5'-tetramethylbenzidine in a mildly acidic buffer. A blue-colored product was produced and turned to yellow after an acidic stop solution was added. The intensity of the color yellow was proportional to the IL-8 amount bound on the plate. The optical density absorbance was measured spectrophotometrically at 450nm in a microplate reader and the concentration of IL-8 was calculated. For the expression of IL-8 concentrations in the samples, a standard curve was used.Optimal threshold values (cut-offs) for biomarkers were determined based on sensitivity and specificity, which were calculated from a ROC curve.
Presepsin amount measurement using ELISA kit | 6 Month - 1 Year
  Presepsin levels were measured in ng/ml using the ELISA method. The measurement procedure was followed according to the manufacturer's instructions. The anti-Presepsin polyclonal antibody was pre-coated on 96-well plates. Blood samples and a biotin-conjugated antibody were added to the wells supplemented with Avidin-Biotin-Peroxidase Complex and 3,3',5,5'-tetramethylbenzidine in a mildly acidic buffer. A blue-colored product was produced and turned to yellow after an acidic stop solution was added. The intensity of the color yellow was proportional to the Presepsin amount bound on the plate. The optical density absorbance was measured spectrophotometrically at 450nm in a microplate reader and the concentration of Presepsin was calculated. For the expression of Presepsin concentrations in the samples, a standard curve was used.Optimal threshold values (cut-offs) for biomarkers were determined based on sensitivity and specificity, which were calculated from a ROC curve.

SECONDARY OUTCOMES:
The Correlation Between Pre-Treatment Pain Presence and Radiographic Success After Pulpotomy Treatment | 1 Year
  The success of treatment was evaluated radiographically after 12 months in teeth with pain related to pre-treatment stimuli.At the end of 12 months; Teeth with no signs of root resorption (internal or external), furcation involvement or periapical radiolucency, no signs of lamina dura loss, and a normal appearance of the periodontal ligament were considered radiographically successful.
The Correlation Between The Severity of Pulp Bleeding During Treatment and Radiographic Success After Pulpotomy Treatment | 1 Year
  The radiographic success of pulpotomy treatment was evaluated at 12 months in teeth with severe pulp bleeding during treatment.At the end of 12 months; Teeth with no signs of root resorption (internal or external), furcation involvement or periapical radiolucency, no signs of lamina dura loss, and a normal appearance of the periodontal ligament were considered radiographically successful.
The Correlation Between Pulp Bleeding Time During Treatment and Radiographic Success After Pulpotomy Treatment | 1 Year
  The radiographic success of pulpotomy treatment was evaluated at the 12th month, depending on the shorter (less than 3 minutes) and longer (3-5 minutes) bleeding duration during treatment.At the end of 12 months; Teeth with no signs of root resorption (internal or external), furcation involvement or periapical radiolucency, no signs of lamina dura loss, and a normal appearance of the periodontal ligament were considered radiographically successful.

CONTACTS AND LOCATIONS:
Overall Officials: AYBİKE BAŞ, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University Faculty of Dentistry, Yakutiye, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahuja S, Surabhi K, Gandhi K, Kapoor R, Malhotra R, Kumar D. Comparative Evaluation of Success of Biodentine and Mineral Trioxide Aggregate with Formocresol as Pulpotomy Medicaments in Primary Molars: An In Vivo Study. Int J Clin Pediatr Dent. 2020 Mar-Apr;13(2):167-173. doi: 10.5005/jp-journals-10005-1740. PMID 32742096
- [Result] Alsanouni M, Bawazir OA. A Randomized Clinical Trial of NeoMTA Plus in Primary Molar Pulpotomies. Pediatr Dent. 2019 Mar 15;41(2):107-111. PMID 30992107
- [Result] Bani M, Aktas N, Cinar C, Odabas ME. The Clinical and Radiographic Success of Primary Molar Pulpotomy Using Biodentine and Mineral Trioxide Aggregate: A 24-Month Randomized Clinical Trial. Pediatr Dent. 2017 Jul 15;39(4):284-288. PMID 29122067
- [Result] Bossu M, Iaculli F, Di Giorgio G, Salucci A, Polimeni A, Di Carlo S. Different Pulp Dressing Materials for the Pulpotomy of Primary Teeth: A Systematic Review of the Literature. J Clin Med. 2020 Mar 19;9(3):838. doi: 10.3390/jcm9030838. PMID 32204501
- [Result] Cordell S, Kratunova E, Marion I, Alrayyes S, Alapati SB. A Randomized Controlled Trial Comparing the Success of Mineral Trioxide Aggregate and Ferric Sulfate as Pulpotomy Medicaments for Primary Molars. J Dent Child (Chic). 2021 May 15;88(2):120-128. PMID 34321144
- [Result] Cuadros-Fernandez C, Lorente Rodriguez AI, Saez-Martinez S, Garcia-Binimelis J, About I, Mercade M. Short-term treatment outcome of pulpotomies in primary molars using mineral trioxide aggregate and Biodentine: a randomized clinical trial. Clin Oral Investig. 2016 Sep;20(7):1639-45. doi: 10.1007/s00784-015-1656-4. Epub 2015 Nov 18. PMID 26578117
- [Result] Donnermeyer D, Dammaschke T, Lipski M, Schafer E. Effectiveness of diagnosing pulpitis: A systematic review. Int Endod J. 2023 Oct;56 Suppl 3:296-325. doi: 10.1111/iej.13762. Epub 2022 May 25. PMID 35536159
- [Result] Elsalhy M, Azizieh F, Raghupathy R. Cytokines as diagnostic markers of pulpal inflammation. Int Endod J. 2013 Jun;46(6):573-80. doi: 10.1111/iej.12030. Epub 2012 Dec 13. PMID 23240887
- [Result] Farges JC, Keller JF, Carrouel F, Durand SH, Romeas A, Bleicher F, Lebecque S, Staquet MJ. Odontoblasts in the dental pulp immune response. J Exp Zool B Mol Dev Evol. 2009 Jul 15;312B(5):425-36. doi: 10.1002/jez.b.21259. PMID 19067439
- [Result] Gonzalez-Lara A, Ruiz-Rodriguez MS, Pierdant-Perez M, Garrocho-Rangel JA, Pozos-Guillen AJ. Zinc Oxide-Eugenol Pulpotomy in Primary Teeth: A 24-Month Follow-up. J Clin Pediatr Dent. 2016;40(2):107-12. doi: 10.17796/1053-4628-40.2.107. PMID 26950810
- [Result] Gopinath VK, Anwar K. Histological evaluation of pulp tissue from second primary molars correlated with clinical and radiographic caries findings. Dent Res J (Isfahan). 2014 Mar;11(2):199-203. PMID 24932190
- [Result] Guo J, Zhang N, Cheng Y. Comparative efficacy of medicaments or techniques for pulpotomy of primary molars: a network meta-analysis. Clin Oral Investig. 2023 Jan;27(1):91-104. doi: 10.1007/s00784-022-04830-1. Epub 2022 Dec 29. PMID 36580161
- [Result] Hirsch V, Wolgin M, Mitronin AV, Kielbassa AM. Inflammatory cytokines in normal and irreversibly inflamed pulps: A systematic review. Arch Oral Biol. 2017 Oct;82:38-46. doi: 10.1016/j.archoralbio.2017.05.008. Epub 2017 Jun 1. PMID 28600966
- [Result] Juneja P, Kulkarni S. Clinical and radiographic comparison of biodentine, mineral trioxide aggregate and formocresol as pulpotomy agents in primary molars. Eur Arch Paediatr Dent. 2017 Aug;18(4):271-278. doi: 10.1007/s40368-017-0299-3. Epub 2017 Aug 5. PMID 28780718
- [Result] Matsuo T, Nakanishi T, Shimizu H, Ebisu S. A clinical study of direct pulp capping applied to carious-exposed pulps. J Endod. 1996 Oct;22(10):551-6. doi: 10.1016/S0099-2399(96)80017-3. PMID 9198445
- [Result] Memar MY, Baghi HB. Presepsin: A promising biomarker for the detection of bacterial infections. Biomed Pharmacother. 2019 Mar;111:649-656. doi: 10.1016/j.biopha.2018.12.124. Epub 2019 Jan 3. PMID 30611989
- [Result] Michaelson PL, Holland GR. Is pulpitis painful? Int Endod J. 2002 Oct;35(10):829-32. doi: 10.1046/j.1365-2591.2002.00579.x. PMID 12406376
- [Result] Ng FK, Messer LB. Mineral trioxide aggregate as a pulpotomy medicament: an evidence-based assessment. Eur Arch Paediatr Dent. 2008 Jun;9(2):58-73. doi: 10.1007/BF03262612. PMID 18534173
- [Result] Ozdemir Y, Kutukculer N, Topaloglu-Ak A, Kose T, Eronat C. Comparative evaluation of pro-inflammatory cytokine levels in pulpotomized primary molars. J Oral Sci. 2015 Jun;57(2):145-50. doi: 10.2334/josnusd.57.145. PMID 26062864
- [Result] Pratima B, Chandan GD, Nidhi T, Nitish I, Sankriti M, Nagaveni S, Shweta S. Postoperative assessment of diode laser zinc oxide eugenol and mineral trioxide aggregate pulpotomy procedures in children: A comparative clinical study. J Indian Soc Pedod Prev Dent. 2018 Jul-Sep;36(3):308-314. doi: 10.4103/JISPPD.JISPPD_1132_17. PMID 30246755
- [Result] Shafaee H, Alirezaie M, Rangrazi A, Bardideh E. Comparison of the success rate of a bioactive dentin substitute with those of other root restoration materials in pulpotomy of primary teeth: Systematic review and meta-analysis. J Am Dent Assoc. 2019 Aug;150(8):676-688. doi: 10.1016/j.adaj.2019.03.002. Epub 2019 Jun 13. PMID 31202439
- [Result] Smail-Faugeron V, Glenny AM, Courson F, Durieux P, Muller-Bolla M, Fron Chabouis H. Pulp treatment for extensive decay in primary teeth. Cochrane Database Syst Rev. 2018 May 31;5(5):CD003220. doi: 10.1002/14651858.CD003220.pub3. PMID 29852056
- [Result] Sorsa T, Gursoy UK, Nwhator S, Hernandez M, Tervahartiala T, Leppilahti J, Gursoy M, Kononen E, Emingil G, Pussinen PJ, Mantyla P. Analysis of matrix metalloproteinases, especially MMP-8, in gingival creviclular fluid, mouthrinse and saliva for monitoring periodontal diseases. Periodontol 2000. 2016 Feb;70(1):142-63. doi: 10.1111/prd.12101. PMID 26662488
- [Result] Stringhini Junior E, Dos Santos MGC, Oliveira LB, Mercade M. MTA and biodentine for primary teeth pulpotomy: a systematic review and meta-analysis of clinical trials. Clin Oral Investig. 2019 Apr;23(4):1967-1976. doi: 10.1007/s00784-018-2616-6. Epub 2018 Sep 20. PMID 30238414
- [Result] Xavier MT, Costa AL, Caramelo FJ, Palma PJ, Ramos JC. Evaluation of the Interfaces between Restorative and Regenerative Biomaterials Used in Vital Pulp Therapy. Materials (Basel). 2021 Sep 3;14(17):5055. doi: 10.3390/ma14175055. PMID 34501145
- [Result] Zehnder M, Delaleu N, Du Y, Bickel M. Cytokine gene expression--part of host defence in pulpitis. Cytokine. 2003 May;22(3-4):84-8. doi: 10.1016/s1043-4666(03)00116-9. PMID 12849707
- [Result] Zou Q, Wen W, Zhang XC. Presepsin as a novel sepsis biomarker. World J Emerg Med. 2014;5(1):16-9. doi: 10.5847/wjem.j.issn.1920-8642.2014.01.002. PMID 25215141
- [Derived] Bas A, Derelioglu SS, Laloglu E. Efficacy of proinflamatory cytokines in the clinical and radiograpic outcomes of different primary molar pulpotomy agents: a comperative randomised study featuring a novel biomarker for pulpal diagnosis. BMC Oral Health. 2024 Oct 15;24(1):1227. doi: 10.1186/s12903-024-04972-6. PMID 39407247